CLINICAL TRIAL: NCT01661543
Title: Substantiating a Health Claim for Pulses (Beans and Peas) and Cholesterol Lowering Abilities
Brief Title: U of A/ U of M Beans and Peas Health Claim Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Innovates Health Solutions (Other); Pulse Canada (Other); University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: QFH-11-044
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — lunatusin, Phaseolus lunatus

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators and data analysts were blinded to participant group assignment.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bean consumption to lower cholesterol (Experimental): This arm will consume 120 grams of cooked beans per day in a food item such as a soup or stew for 5 out of 7 days for 6 weeks.
  The bases (i.e. vegetables, broth, seasonings, etc) for all food items are the same in all groups.
  Interventions: Dietary Supplement: Beans
- Control (rice) consumed to show results (Placebo Comparator): The control group will consume 110 grams (~3/4 c) of rice per day in a food item such as a soup or study for 5 out of 7 days for 6 weeks. This amount of rice is similar in volume to 120g of beans or peas.
  The bases (i.e. vegetables, broth, seasonings, etc) for all food items are the same in all groups.
  Interventions: Dietary Supplement: Control (rice)
- Peas consumed to lower cholesterol (Experimental): This arm will consume 120 g of cooked peas per day per day in a food item such as a soup or stew for 5 days out of 7 days for 6 weeks.
  The bases (i.e. vegetables, broth, seasonings, etc) for all food items are the same in all groups.
  Interventions: Dietary Supplement: Peas

INTERVENTIONS:
Dietary Supplement: Beans — 120g of beans per day for 5 out of 7 days per week will be given to participants for 6 weeks to determine the cholesterol lowering effects of various pulses.
  Arms: Bean consumption to lower cholesterol
Dietary Supplement: Control (rice) — 110g (3/4 c) of rice per day will be given to the control group to demonstrate the cholesterol lowering effects of the experimental group. This amount of rice equates to a similar volume as 120g of cooked beans or peas.
  Arms: Control (rice) consumed to show results
Dietary Supplement: Peas — 120 grams of peas will be consumed 5 out of 7 days per week
  Arms: Peas consumed to lower cholesterol

SUMMARY:
The purpose of this study is to compare how regularly eating (dried, cooked) beans or peas or rice (control) contained in foods (such as stews or soups) lowers blood lipids, particularly Low Density Lipoprotein cholesterol (LDL-c) in adult men and women with mildly elevated LDL-c . The investigators hypothesize that regularly eating beans or peas will significantly improve LDL-c in these people.

Participants in this study will consume 1 study food item, 5 out of 7 days per week containing beans or peas or rice for a total of 6 weeks. Measuring changes in blood and urinary polyphenol levels may help to verify whether these ingredients play a role in the beneficial actions attributed to regularly eating pulses. It may subsequently assist with the identification of the beneficial bean/pea components. This study will could benefit people who wish to incorporate beans and/or peas into their diet. It may also benefit Canadian pulse growers by enhancing development of food products for human consumption and supporting marketing strategies to increase awareness that a diet rich in pulses can improve LDL-c. This in turn, could enable crop breeders to select for plants that are rich in these compounds.

DETAILED DESCRIPTION:
OBJECTIVES: The aim of this study is to conduct a multi-centre randomized, controlled trial to compare the biological effectiveness of bean vs rice and peas vs rice (control) on LDL-cholesterol after 6 weeks in mildly hypercholesterolemic men and women. The primary outcome is LDL-cholesterol at 6 weeks, adjusted for baseline.

In addition, the effects of beans and peas on other factors associated with cardiovascular disease. Secondary outcomes are: total cholesterol, triglycerides, high density lipoprotein-cholesterol, non-HDL cholesterol, body weight, body mass index, glucose, insulin, glycated hemoglobin and biomarkers of vascular function; these are measured at 3 and 6 weeks. LDL-cholesterol at 3 weeks is also a secondary outcome. Inflammation and metabolism will be investigated. Participants' assessment of study food acceptability, satiety and gastrointestinal responses will also be collected.

BACKGROUND: Pulses (beans, peas, lentils and chickpeas) are healthy foods that contain twice the amount of protein as cereals, are very high in fibre, key vitamins and minerals like folate and iron and are low in fat. Canada is the world's largest producer and exporter of lentils and peas, and Alberta produced 34% of the pea crop and 12% of beans in 2010. Current consumption of pulses in Canada is low, due to a lack of pulse-based convenient food products. An approved health claim can drive interest in development of food products with particular ingredients as seen with oat beta-glucan. Experts agree that existing evidence for the cholesterol-lowering effects of pulses is particularly strong for beans, but more studies are needed to show the effects of peas, lentils and chickpeas are comparable to beans. Results from this study will be used to substantiate a health claim for beans and other pulse crops in the future, similar to the health claims that exist for beta-glucan and plant sterols.

METHODS AND PROCEDURES: This multi-center study will compare the effects of consuming beans (pinto, black, Great Northern, navy) to control (rice-based) and peas (yellow, green) to control (rice-based) foods for 6 weeks on Low Density Lipoprotein-Cholesterol in mildly hypercholesterolemic (>3 mmol/L and < 5mmol/L; not on medications) adults. There will be 3 study arms: i) beans, ii) peas, and iii) rice (control). The study groups will be asked to consume food items containing 120 grams of cooked beans or cooked peas daily for 6 weeks. The control group will be asked to consume 110 g of cooked, convert rice (one 3/4 cup serving per day) foods in matrices identical to those containing beans or peas for 6 weeks. The study or control foods will be incorporated into the participants normal dietary pattern. All food items will be provided to participants free of charge. Food items, generally in the form of soups or stews, will be developed by a collaborator in Food Science at the University of Manitoba in the initial phase of this project .

The investigators plan to recruit approximately 180 participants (n= 75 participants at the University of Manitoba and n= 105 at University of Alberta). Interested individuals (potential participants) will first attend a screening visit. The screening visit procedures will be discussed prior to the screening visit, including the need to fast (i.e., no food or beverage intake except water for 12 hours) for blood sampling to determine if Low-density-lipoprotein-cholesterol and triglyceride levels are within acceptable range. Once at the screening visit, individuals will be provided with a description of the study by the investigating team's study coordinator. The eligibility criteria will be reviewed with candidates by the investigating team's study coordinator to assess their suitability for the study. Individuals meeting all inclusion/exclusion criteria will be contacted by the study coordinator with this information. All individuals who are screened will be contacted by the study coordinator once eligibility has been confirmed. An appointment for a baseline assessment meeting will be scheduled for those who are eligible and who confirm interest in the study; those who are not eligible or who are eligible and no longer wish to participate will be thanked for their time.

At the baseline assessment visit individuals will be reminded of the study description and will be asked to provide written informed consent at this time.

Once enrolled, participants will undergo a complete medical history including age, sex, alcohol use, exercise habits, current medical problems, medication and family history of previous events such as stroke and diabetes. A fasting blood sample will be obtained to assess plasma lipid profile.

Participants will be asked to attend 4 in-person clinic visits over the duration of the study for screening, baseline assessment, and at 3 and 6 weeks (at the end of the study).

Once identified and after giving informed consent, participants will be randomized to one of the 3 study arms. The randomization will be either computer generated, or done manually by a study coordinator for both sites. Each participant will be given a randomized number, and will be used for all study documentation.

Participants will fill out questionnaire relating to demographics, lifestyle, food intake, gastrointestinal responses etc.

The baseline visit will include a height and weight measurement and waist circumference. Blood pressure will be recorded. Participants medications and current medical conditions will be documents. The three day food record (completed at home) will be collected. Fasting blood sample will be drawn for lipid profile assessment (LDL-c, total cholesterol, triglycerides, HDL-cholesterol, non-HDL cholesterol), insulin, glucose, glycated hemoglobin, polyphenols and biomarkers of vascular function, inflammation and metabolism. Blood required will not exceed 60mL.

Randomization will be done at the baseline visit. Prior to leaving, participants will be provided with the first 3-week supply of assigned foods and instruction about how to prepare and consume them, and will be reminded to fast before their next visit. This visit will take approximately 2.5 hours.

Week 3 visit: height, weight and waist circumference measurements. Blood pressure will be recorded. Participants will be assessed for changes in their medications and current medical conditions. The 3 day food record (completed at home) will be collected. Urine sample will be collected. A fasting blood sample will be drawn for assessment of lipid profile, insulin, glucose, glycated hemoglobin, polyphenols and biomarkers of vascular function, inflammation and metabolism. The total blood required will not exceed 60mL.

Participants will complete a questionnaire to assess compliance, acceptability of the study foods, satiety, GI responses and any adverse events. Questions will be addressed. Before leaving, participants will be provided with the second 3-week supply of assigned foods, and instructions about how to prepare and consume them. Participants will be reminded to fast prior to next visit. Visit will take approximately 2 hours.

Week 6 visit: Measurements taken for height, weight and waist circumference, and blood pressure will be repeated. Participants will be assessed for changes in medications and current medical conditions. Urine sample will be collected for polyphenols. A fasting blood sample will be drawn for assessment of primary outcome, LDL-c, along with the rest of the lipid measures (see above), insulin, glucose, glycated hemoglobin, polyphenols, and biomarkers of vascular function (University of Manitoba only), inflammation and metabolism. Total blood will not exceed 60 mL.

Participants will complete a questionnaire to assess compliance, acceptability of the foods, satiety, Gastrointestinal responses and any adverse events. Total time required, approximately 2.5 hours. Completion of this visit marks the end of the study. Participants will be paid, and thanked for their time.

ELIGIBILITY:
Inclusion Criteria:

* Male, or non-pregnant, non-lactating females, aged 20 to 75 years; This age range allows for a large variety of participants.
* LDL-cholesterol >3.00 mmol/L and <5.00 mmol/L; Cholesterol is high enough that a lowering can be seen, but low enough that the participant is not taking medications or alternative measures to lower cholesterol.
* Fasting triglycerides <4.00 mmol/L; Low enough that it is not dangerous to participant, but high enough to see a lowering effect.
* Stable body weight (±5%) for the past 3 months and BMI of 20-40; Participants with high BMI are more likely to have high lipid levels, it is important to have a stable body weight so energy requirements are not drastically changing during the study period.
* Must be on a stable regime for the past 3 months if taking medications or if taking vitamin and mineral/dietary/herbal supplements; Stable regime reduces risk of any changes during study.
* Able to read, write and communicate orally in English; All questionnaires and communication will be completed in English.

Willing to comply with the protocol requirements, including a stable level of physical activity during the study and no other pulse-containing foods consumed during the study; this will ensure the most valid results.

Willing to provide informed consent.

Exclusion Criteria:

* Regular high pulse consumption (>2 servings per week); Any additional pulse consumption will affect the outcome of the study.
* Use of medications to lower blood lipids or to lower blood glucose; the aim of the study is to prove the cholesterol lowering capabilities of beans and peas, any other methods of blood lipid lowering will skew data.
* Use of non-prescription products designed to lower blood lipids (e.g. margarine or yogurt with added plant sterols) within the past 3 months; see above
* Medical history of liver disease, renal insufficiency, inflammatory bowel disease or other gastrointestinal disorders influencing gastrointestinal motility or nutrient absorption; this will decrease effectiveness of bean/ consumption.
* Any active medical or surgical condition(s) within the past 3 months precluding study participation; participants must be in a stable condition with no recovery or pending surgery.
* Conditions or medications which are likely to increase the risk to the participants or study personnel, or to reduce the ability of the participant to comply with the protocol, or affect the results;
* History of gastrointestinal reactions or allergies to beans, peas or rice-based foods, or to one or more ingredients in the study foods which significantly limits the number of study foods that can be consumed.
* Currently participating in or having participated in a food intervention study within the last 3 months.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Fasting Low Density Lipoprotein-cholesterol (LDL-c) at 6 weeks | 6 weeks
  Fasting LDL-c at 6 weeks

SECONDARY OUTCOMES:
Fasting LDL-cholesterol at 3 weeks | 3 weeks
  Fasting LDL-cholesterol at 3 weeks
Fasting HDL-cholesterol | 3 and 6 weeks
  Fasting HDL-cholesterol at 3 and 6 weeks
Fasting non-HDL-cholesterol | 3 and 6 weeks
  Fasting non-HDL-cholesterol at 3 and 6 weeks
Fasting Total Cholesterol | 3 and 6 weeks.
  Fasting total cholesterol at 3 and 6 weeks
Fasting Triglycerides | 3 and 6 weeks
  Fasting triglycerides at 3 and 6 weeks
Glycated hemoglobin | 3 and 6 weeks
  Hb-A1c at 3 and 6 weeks
Fasting Glucose | 3 and 6 weeks
  Fasting glucose at 3 and 6 weeks
Fasting Insulin | 3 and 6 weeks
  Fasting insulin at 3 and 6 weeks
Systolic Blood Pressure | 3 and 6 weeks
  Systolic blood pressure at 3 and 6 weeks
Diastolic Blood Pressure | 3 and 6 weeks
  Diastolic blood pressure at 3 and 6 weeks
Body weight | 3 and 6 weeks
  Body weight at 3 and 6 weeks
Waist circumference | 3 and 6 weeks
  waist circumference at 3 and 6 weeks
Hip circumference | 3 and 6 weeks
  Hip circumference at 3 and 6 weeks
Body Mass Index (BMI) | 3 and 6 weeks
  BMI (weight/height*height) at 3 and 6 weeks

OTHER OUTCOMES:
Dietary Intake from 3-day Food Records | 1, 3 and 6 weeks
  Energy, macronutrient and micronutrient calculated from 3-day food records collected during weeks 1, 3 and 6
Satiety | 1, 3 and 6 weeks
  There are no standarized protocols or questionnaires to measure satiety. Satiety will be calculated from participant self-reports of the following questions and responses will be recorded on a 100 mm analogue cale). Q1 How hungry to you feel; Reponses 0=No hungry at all; 100=have never been more hungry; Q2 How satisfied do you feel? Responses0 0=I am completely empty, 100=I cannot eat another bite; Q3 How full do you feel? Responses 0=Not full at all, 100=Totally full; Q4 How much more do you think you can eat? Responses 0=Nothing at all, 100=A lot. These questions will be answered 30 mins after consuming 1 of the study foods during weeks 1, 3 and 6.
Changes in GI function | 1, 3 and 6 weeks
  There are no standarized questionnaires about gastrointestinal function. Q1 Any changes in flatulence (gas) over the past week? No/Yes. If yes: has frequency increased or decreased? Increased/Decreased; rate amount of change, scale 1-5, 1=little change 5=lot of change. Q2: Any changes in stool frequency over past week? No change/ increased/ decreased. If changed, rate amount of change, scale 1-5, 1=little change 5= lot of change; Q3: Changes in stool consistency, such as stool softer/looser or harder/firmer? No/yes; if yes, is stool softer or harder? Rate change in stool consistency, scale 1-5, 1=little, 5=a lot of change; Q4. Have you felt bloating during the past week? No/yes. Rate amount of change in bloating, scale 1-5, 1=little change, 5=lot of change. Q5 Were any of your normal daily activities affected during the past week by: (check all that apply): Flatulence, stool frequency, stool consistency, bloating, no changes to normal daily activities
Adverse Events | 3 and 6 weeks.
  Questions about any adverse events experienced during trial, weeks 3 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda C Bell, PhD, Principal Investigator — University of Alberta; Linda McCargar, PhD, Study Chair — University of Alberta; Cathy Chan, PhD, Study Chair — university; Spencer Proctor, PhD, Study Chair — University of Alberta; Jocelyn Ozga, PhD, Study Chair — University of Alberta; David Wishart, PhD, Study Chair — University of Alberta; Carla Taylor, PhD, Study Chair — University of Manitoba; Peter Zahradka, PhD, Study Chair — University of Manitoba; Michel Aliani, PhD, Study Chair — University of Manitoba
Locations (2):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - University of Manitoba, Winnipeg, Manitoba

REFERENCES:
- [Derived] Bell RC, Zahradka P, Aliani M, Liang Y, Jarman M, MacKenzie M, Chan C, Ozga J, Proctor S, Wishart D, Taylor CG. A Comparison of Dry Bean and Pea Consumption on Serum Cholesterol: A Randomized Controlled Trial in Adults with Mild Hypercholesterolemia. J Nutr. 2024 Nov;154(11):3375-3387. doi: 10.1016/j.tjnut.2024.09.011. Epub 2024 Sep 30. PMID 39357673
- [Derived] Pauls SD, Du Y, Clair L, Winter T, Aukema HM, Taylor CG, Zahradka P. Impact of Age, Menopause, and Obesity on Oxylipins Linked to Vascular Health. Arterioscler Thromb Vasc Biol. 2021 Feb;41(2):883-897. doi: 10.1161/ATVBAHA.120.315133. Epub 2020 Dec 31. PMID 33380172